CLINICAL TRIAL: NCT02326246
Title: Multi-parametric Magnetic Resonans Imaging in the Diagnosis and Surveillance of Low-risk Prostate Cancer
Brief Title: MRI in Active Surveillance of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Maria C Elkjær, MD, ph.d. student, Aarhus University Hospital Skejby
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U-Aarhus
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: MRI; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- men with low-risk PC (Experimental): men newly diagnosed with low-risk prostate cancer and put in an active surveillance (AS) program. Eight weeks post TRUS-guided biopsies they are scanned with a multi-parametric magnetic resonans imaging (mMRI). If the scans shows a PIRADS 4 or 5 lesion, MRI-guided biopsies are performed. Otherwise the patients will continue in the AS program as usual. The mMRI will in these cases be repeated after 1 year.
  Interventions: Other: multi-parametic MRI

INTERVENTIONS:
Other: multi-parametic MRI

SUMMARY:
The purpose of this study is to investigate the hypothesis, that mMRI provides a more accurate and secure interpretation of the aggressiveness of prostate cancer initially/before mMRI defined as low risk. In doing so we will investigate and assess the affect of mMRI on gleason score upgrade, risk classification upgrade and changes in treatment strategy (active surveillance vs. operation).

DETAILED DESCRIPTION:
At the urological department K, Aarhus University Hospital (AUH), approx. 500 TRUS biopsies are performed each year and about 125 intermediate/high risk patients undergo radical prostatectomy (RP). At any time approx. 50 men with low-risk PC is in active surveillance (AS).

The MRIs will all be performed with a 3 Tesla MRI system with a phased-array coil including standard T1 and T2-weighted sequences, diffusion-weighted sequences with different b-values and a dynamic contrast sequence of the prostate gland. In patients in whom a previous mMRI has shown tumor, the MRGBs will be performed with the commercially available DynaCAD-equipment designed for in-bore MR-guided prostate biopsies.

The Study Design: a prospective study of 60* patients enrolled in an AS program. From late 2014 and approximately one year forward, all patients put in active surveillance after the diagnosis of low risk PC, will after that decision be offered an additional mMRI scan.

If the mMRI gives rise to suspicion of significant cancer, MRGB will be taken. Results of these biopsies will be assessed, and in some cases gleason score will be up-grated, risk classification will be up-grated and the decision to keep the patient in AS will have to be changed, and active treatment will be recommended. If the scan finds no reason to change strategy, the patient will have the usual follow-ups in the clinic, which in an AS program usually consists of control PSA value every 3 months, and new TRUS guided biopsies after 12 months or if PSA rises. Parallel to the usual control program we will perform a new mMRI once a year to assess if there is any progression in the disease, and again do MRGB if this is the case.

The study will require access to the patient journals. We will look at patient demographics, specification on the PC found, histology and blood samples.

In the study we will consult a statistician as the work progresses, to ensure the quality of our data work and conclusions.

Recruitment of participants and obtaining informed consent At the department's weekly multi-disciplinary conference (MDT), the tissue samples, taken by ultrasound, are presented. On this conference future treatment strategy for each patient is planned. At this conference it will be possible to identify possible candidates for the project. Afterwards, when the patient receives the answer in the out patient clinic, by a hospital doctor, he will be offered an interview with the study responsible Ph.D. student. The patient is offered to bring a companion to the conversation, that can occur on the same day or later, depending on the patient's preference and the opportunity to be escorted. At this conversation, oral and written information is given in a suitable consultation room in the outpatient clinic, and it will be evaluated if the patient is suitable for inclusion. The patient is offered 24 hours to think. The written consent is obtained when the patient indicates not having a need for further information and reflection.

Inclusion is expected to commence in late year2014, when permission is granted from the Ethics Committee. Expectedly the inclusion of patients will be completed within 12 months and thus expected to end late of year 2015.

Side effects, risks and drawbacks The same precautions on MRI safety will be taken as with other clinical patients using the existing metal table, and therefore there are no known risks associated with the actual scan. While completing the scan intravenous gadolinium-containing contrast is used. This is excreted through the kidneys and is safe for patients with normal renal function (see exclusion criteria). The most common side effects of the proposed contrast agent Dotarem® include: a feeling of heat, cold and / or pain at the injection site and transient headache and tingling sensations in the skin (more than 1 out of 10 individuals). The patient may develop an allergic reaction to the contrast, and in the most serious cases the is a risk of heart failure, slow heartbeat, irregular heartbeat, respiratory, mucosal swelling in the throat and pleuritis in the lungs, constriction of the airways, breathlessness and sneezing. This is very rare (less than 1 in 10 000 individuals). An allergic reaction will be immediately treated according to current guidelines in the department. The patient will be questioned to known allergy to MRI contrast agent both be inclusion, and immediately before the injection.

In cases where we find a basis for further tissue samples from the MRI, there will be a risk of sepsis and bleeding in the rectum. This risk is assessed to be far lower than by the usual use TRUS samples, as there usually will only be 2-4 tissue samples as compared to 12 by the usual method. Patients will receive preventive antibiotics as usually given with TRUS (ciprofloxacin). In addition, the selection can be associated with discomfort / pain. This is expected to be less than with the usual procedure, as there usually will be fewer biopsies taken.

Patients with prostate cancer are currently not routinely examined with MR imaging before surgery. Patients who agree to participate in the trial will thus have a scan they would not otherwise have received. Participation in the study, therefore, means that the patient must visit the hospital a second time. If MRI guided tissue samples must be taken it will also mean one or two extra trips to the hospital (depending on the histology).

Practical and economical aspects The study is planned to be performed at Department of Urology K and the department of MRI, Aarhus University Hospital - Skejby, to commence September 1th 2014 and continue for three years forward.

The project is partly financed by the Danish cancer research foundation. Patients will not receive remuneration.

* (The no. of patients is estimated by a power analysis based on numbers found from two other relevant studies on AS and mMRI in PC. Having an α-value = 0.05 and a β-value of 0.8 gives a minimum of 47 patients in the group. Expecting there will be some variations this is adjusted by including 60 patients in the group.)

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* PC and put in AC,
* No contraindications to MRI,
* Written informed consent

Exclusion Criteria:

* Lack of ability to consent,
* Non-MRI compatible metal in the body,
* Claustrophobia,
* Heavy obesity (largest circumference more than 180 cm),
* Moderate/severe kidney malfunction
* Known allergy to MRI contrast

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
gleason up-grate | 1 year

SECONDARY OUTCOMES:
changes in the treatment strategy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Elkjær, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus N, Denmark